CLINICAL TRIAL: NCT01392482
Title: IBIS: Italian Burden of Illness on Schizophrenia & Bipolar Disorder
Acronym: IBIS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-NIT-XXX-2011/1
Record Dates: First submitted 2011-06-29; First posted 2011-07-12 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Schizophrenia; Bipolar Disorder
Keywords: Schizophrenia; Bipolar Disorder
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- treatment with antipsychotics: 40 LHU covering about 18 millions inhabitants distributed all over Italy with a coverage of nearly 100% of Italian regions. All subjects will be included in the analysis who have received treatment with antipsychotics (typical and / or atypical) between January 1, 2009 and June 30, 2010 and diagnosed with schizophrenia and / or Bipolar Disorder.

SUMMARY:
Multicentre, retrospective observational cohort study based on LHU administrative databases aimed to described the pharmacoutilization of antipsychotics in patients affected by schizophrenia and bipolar disorder, the resource consumption and medication adherence. A sub analysis will be performed for those patients switching from Quetiapine IR to Quetiapine XR and comparing the periods before and after the switch.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Schizophrenia or BD (appendix for ICD9-10 codes) or an antipsychotic prescription during the period 1/1/2009-30/06/2010
* patients must be assisted in the LHU for the year before the enrollment ( period 1/1/2009-30/06/2010) until 31/12/2010 or death date if earlier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients from 40 LHU
Sampling Method: Non-Probability Sample
Enrollment: 751725 (Actual)
Dates: Start 2011-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Describe the pharmacoutilization of antipsychotics treatment (including typical and atypical) for patients affected by schizophrenia and bipolar disorder in order to evaluate the level of treatment variability for these patients | Index Data up to 18 months
  The reference date, the Index Date for patients included in the analysis will be identified on the basis of the date of first prescription of antipsychotics in the period January 1, 2009 - June 30, 2010 or, for those that do not result in treatment with antipsychotics, according to the date of diagnosis of schizophrenia or bipolar disorder, if that date is within the period 1 January 2009 - June 30, 2010, otherwise the date will be January 1, 2009

SECONDARY OUTCOMES:
Describe the costs of illness of patients with schizophrenia or bipolar disorder | Index Data up to 18 months
  The reference date, the Index Date for patients included in the analysis will be identified on the basis of the date of first prescription of antipsychotics in the period January 1, 2009 - June 30, 2010 or, for those that do not result in treatment with antipsychotics, according to the date of diagnosis of schizophrenia or bipolar disorder, if that date is within the period 1 January 2009 - June 30, 2010, otherwise the date will be January 1, 2009
To evaluate adherence level for patients treated with antipsychotics | Index Data up to 18 months
  The reference date, the Index Date for patients included in the analysis will be identified on the basis of the date of first prescription of antipsychotics in the period January 1, 2009 - June 30, 2010 or, for those that do not result in treatment with antipsychotics, according to the date of diagnosis of schizophrenia or bipolar disorder, if that date is within the period 1 January 2009 - June 30, 2010, otherwise the date will be January 1, 2009
A sub analysis will be performed to evaluate any differences in terms of cost of illness and medication adherence for those patients switching from quetiapine IR to quetiapine XR in order to understand the implications of the different formulations. | Index Data up to 18 months
  The reference date, the Index Date for patients included in the analysis will be identified on the basis of the date of first prescription of antipsychotics in the period January 1, 2009 - June 30, 2010 or, for those that do not result in treatment with antipsychotics, according to the date of diagnosis of schizophrenia or bipolar disorder, if that date is within the period 1 January 2009 - June 30, 2010, otherwise the date will be January 1, 2009

CONTACTS AND LOCATIONS:
Overall Officials: Flore La Tour, Study Chair — AstraZeneca; Raffaele Sabia, Study Director — AstraZeneca
Locations (16):
- Italy (16):
  - Research Site, Arezzo, AR
  - Research Site, Bergamo, BG
  - Research Site, Bolzano, BZ
  - Research Site, Forlì, FC
  - Research Site, Ferrara, FE
  - Research Site, Florence, FI
  - Research Site, Lecce, LE
  - Research Site, Matera, MT
  - Research Site, Monza E Brianza, MZ
  - Research Site, Piacenza, PC
  - Research Site, Ravenna, RA
  - Research Site, Ragusa, RG
  - Research Site, Teramo, TE
  - Research Site, Milan
  - Research Site, Molise
  - Research Site, Rome

REFERENCES:
- [Background] Brown S. Excess mortality of schizophrenia. A meta-analysis. Br J Psychiatry. 1997 Dec;171:502-8. doi: 10.1192/bjp.171.6.502. PMID 9519087
- [Background] Tabbane K, Joober R, Spadone C, Poirier MF, Olie JP. [Mortality and cause of death in schizophrenia. Review of the literature]. Encephale. 1993 Jan-Feb;19(1):23-8. French. PMID 8275890
- [Background] Opler LA, Caton CL, Shrout P, Dominguez B, Kass FI. Symptom profiles and homelessness in schizophrenia. J Nerv Ment Dis. 1994 Mar;182(3):174-8. doi: 10.1097/00005053-199403000-00008. PMID 7906710
- [Background] Begley CE, Annegers JF, Swann AC, Lewis C, Coan S, Schnapp WB, Bryant-Comstock L. The lifetime cost of bipolar disorder in the US: an estimate for new cases in 1998. Pharmacoeconomics. 2001;19(5 Pt 1):483-95. doi: 10.2165/00019053-200119050-00004. PMID 11465308
- [Background] Foster RH, Goa KL. Risperidone. A pharmacoeconomic review of its use in schizophrenia. Pharmacoeconomics. 1998 Jul;14(1):97-133. doi: 10.2165/00019053-199814010-00009. PMID 10182198
- [Background] Keller MB, Lavori PW, Klerman GL, Andreasen NC, Endicott J, Coryell W, Fawcett J, Rice JP, Hirschfeld RM. Low levels and lack of predictors of somatotherapy and psychotherapy received by depressed patients. Arch Gen Psychiatry. 1986 May;43(5):458-66. doi: 10.1001/archpsyc.1986.01800050064007. PMID 3083800
- [Background] Kendler KS, Gallagher TJ, Abelson JM, Kessler RC. Lifetime prevalence, demographic risk factors, and diagnostic validity of nonaffective psychosis as assessed in a US community sample. The National Comorbidity Survey. Arch Gen Psychiatry. 1996 Nov;53(11):1022-31. doi: 10.1001/archpsyc.1996.01830110060007. PMID 8911225
- [Background] Tondo L, Baldessarini RJ. Reduced suicide risk during lithium maintenance treatment. J Clin Psychiatry. 2000;61 Suppl 9:97-104. PMID 10826667
- [Background] Kelly GR, Scott JE, Mamon J. Medication compliance and health education among outpatients with chronic mental disorders. Med Care. 1990 Dec;28(12):1181-97. doi: 10.1097/00005650-199012000-00006. PMID 2250501
- [Background] Duncan JC, Rogers R. Medication compliance in patients with chronic schizophrenia: implications for the community management of mentally disordered offenders. J Forensic Sci. 1998 Nov;43(6):1133-7. PMID 9846389
- [Background] The Scottish First Episode Schizophrenia Study. II. Treatment: pimozide versus flupenthixol. The Scottish Schizophrenia Research Group. Br J Psychiatry. 1987 Mar;150:334-8. doi: 10.1192/bjp.150.3.334. PMID 2889495
- [Background] Young JL, Zonana HV, Shepler L. Medication noncompliance in schizophrenia: codification and update. Bull Am Acad Psychiatry Law. 1986;14(2):105-22. PMID 2873851
- [Background] Buchanan A. A two-year prospective study of treatment compliance in patients with schizophrenia. Psychol Med. 1992 Aug;22(3):787-97. doi: 10.1017/s0033291700038228. PMID 1357703
- [Background] Keck PE Jr, McElroy SL, Strakowski SM, West SA, Sax KW, Hawkins JM, Bourne ML, Haggard P. 12-month outcome of patients with bipolar disorder following hospitalization for a manic or mixed episode. Am J Psychiatry. 1998 May;155(5):646-52. doi: 10.1176/ajp.155.5.646. PMID 9585716
- [Background] Catalan VS, LeLorier J. Predictors of long-term persistence on statins in a subsidized clinical population. Value Health. 2000 Nov-Dec;3(6):417-26. doi: 10.1046/j.1524-4733.2000.36006.x. PMID 16464201
- [Background] Weiden PJ, Kozma C, Grogg A, Locklear J. Partial compliance and risk of rehospitalization among California Medicaid patients with schizophrenia. Psychiatr Serv. 2004 Aug;55(8):886-91. doi: 10.1176/appi.ps.55.8.886. PMID 15292538
- [Derived] Degli Esposti L, Sangiorgi D, Mencacci C, Spina E, Pasina C, Alacqua M, la Tour F. Pharmaco-utilisation and related costs of drugs used to treat schizophrenia and bipolar disorder in Italy: the IBIS study. BMC Psychiatry. 2014 Oct 14;14:282. doi: 10.1186/s12888-014-0282-z. PMID 25312446